CLINICAL TRIAL: NCT01663571
Title: STAT3 in T Cells: At The Crossroads of Inflammation and Cancer
Status: Terminated | Type: Observational
Why Stopped: Study is permanently closed to enrollment .Collection of private identifiable information is complete Analysis of private identifiable information is complete
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 11-01293
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsy specimens from cutaneous T cell lymphoma (CTCL) patients and benign skin conditions namely eczema, dermatitis and psoriasis will be obtained through a standard punch biopsy procedure from the skin lesion. The investigators will assay the mRNA levels of the transcription factors of the different T effector cells by qPCR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Protocol Summary

Constitutive STAT3 activity is implicated in many malignancies including Cutaneous T Cell Lymphoma. It is also essential for Th17 differentiation, a subset of CD4 effector T cell, implicated in chronic inflammatory conditions and possibly CTCL. HDAC inhibitors have shown activity in CTCL but their exact mechanism of action is not known. It is known that HDAC inhibitors regulate STAT3 transcriptional activity and hence can potentially be active in CTCL through modulation of the STAT3 pathway. The hypothesis is that Th17 cytokines contribute to the initiation of cancer by creating a pro-inflammatory microenvironment that predisposes cells to neoplastic transformation. To probe this, the investigators will compare the differences in cytokine production and gene expression in the skin resident T cells from patients with benign dermatoses and CTCL as well as in the blood/circulating lymphocytes of healthy donors and Sezary syndrome (SS). The investigators will also investigate whether HDAC inhibitors have a direct impact on the number of Th17 cells, the cytokine production by these cells and phosphorylated STAT3 protein in CTCL with subsequent treatment cycles.

The objectives of this study are 1. Observe the epigenetic, transcriptional and phenotypic changes that take place in T cell during malignant transformation 2. Understand the mechanism of action of HDAC inhibitors in CTCL.

Methods: Skin biopsy specimens from cutaneous T cell lymphoma (CTCL) patients and benign skin conditions namely eczema, dermatitis and psoriasis will be obtained through a standard punch biopsy procedure from the skin lesion.

Additionally, 15 ml of peripheral blood from CTCL patients who have Sezary syndrome (SS) and from patients with benign skin condition will be collected.

CTCL patients, who are starting treatment with HDAC Inhibitors namely Vorinostat and Romidepsin, will have a total of 3 skin biopsies and/or blood draws. The first procedure would be before starting treatment with either of these HDAC inhibitors. Two more skin biopsies and/or blood draws will be performed after first and second cycle of treatment.

Levels of Th17 cytokines, IL-17, IL -22 and pSTAT3 protein will be determined by IHC staining in the skin and cytokine levels in the blood will be assayed by sandwich ELISA method.The investigators will also assay the mRNA levels of the transcription factors of the different T effector cells by qPCR.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with CTCL that are starting new form of treatment and adult patients with benign dermatoses.

Exclusion Criteria:

* patients with lymphomas other than CTCL or leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Cutaneous T cell Lymphoma (CTCL), either newly diagnosed or with progression of disease. Patients with Eczema, psoriasis and dermatitis are also eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
Measure the levels of Th 17 cytokines namely Il-17 and Il-22 in CTCL | 2 -3 years

SECONDARY OUTCOMES:
Identify STAT3 mutations in CTCL | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Koralov, PhD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States